CLINICAL TRIAL: NCT02560415
Title: Patient-centric Model for Remote Management, Treatment and Rehabilitation of Children With Autism - Michelangelo / GOLIAH (Gaming Open Library for Intervention in Autism at Home) Project
Brief Title: Gaming Open Library for Intervention in Autism at Home (GOLIAH /MICHELANGELO)
Acronym: MICHELANGELO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDRCB2014-A-00170-47 - P120914; EU: FP7-ICT-2011-7 (n°288241) (Other Grant/Funding Number: ERNB: 140190-31)
Record Dates: First submitted 2015-09-21; First posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Serious Game; Controlled trial; Denver model
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Experimental (Experimental): Gaming Open Library for Intervention in Autism at Home plus Treatment as usual
  Interventions: Device: Experimental; Behavioral: Comparator
- 2: Comparator (Active Comparator): Treatment as usual
  Interventions: Behavioral: Comparator

INTERVENTIONS:
Device: Experimental — Gaming Open Library for Intervention in Autism at Home plus Treatment as usual
  Arms: 1: Experimental
Behavioral: Comparator — Treatment as usual

SUMMARY:
To meet the required intensive intervention hour for treating children with autism spectrum disorder (ASD), the investigators developed an automated serious gaming platform (11 games) to deliver intensive intervention at home (GOLIAH). The major objective of the study is to test GOLIAH during a 6-month matched controlled exploratory study were to assess (1) the usefulness and acceptability of the gaming platform; (2) how experimental children performed using the different Imitation and JA games; and (3) whether children from the experimental group improved significantly more than children treated as usual (control group).

DETAILED DESCRIPTION:
Background: To meet the required intensive intervention hour for treating children with autism spectrum disorder (ASD), the investigators developed an automated serious gaming platform (11 games) to deliver intensive intervention at home (GOLIAH) by mapping the Imitation and Joint Attention (JA) subset of age-adapted stimuli from the Early Start Denver Model (ESDM) intervention. For the purpose of this study, 24 ASD children will be recruited (one half in Pisa and the other half in Paris). They will be divided into two groups: an Experimental group (N=14) and a Control group (N=10). The Control group will not go through the training sessions, they will participate only in the assessment sessions. All patients will be referred to treatment as usual, according to local facilities.

The protocol is organized into 3 periods (with two assessments at T0 and T6).

* During the initial stage of the protocol (T0), all the ASD children (experimental participants and controls) will be evaluated during a clinical session.
* During the rehabilitation period, only half of the children will participate in the training sessions designed to improve their imitation and joint attention capacities.
* During the final stage of the protocol (T6), all children will be evaluated again during a second clinical session.

The clinical assessments will occur at stage 0 and at stage 6. The same tools will be used for these two assessments. The improvement of children's capabilities will be measured by the progress made between stage 0 and stage 6. The investigators will be able to affirm that the training was beneficial by comparing the clinical session performance between the trained and control children.

ELIGIBILITY:
Inclusion Criteria:

* a current diagnosis of ASD confirmed by clinical assessment and the Autism Diagnostic Interview-Revised;
* an intellectual quotient ≥ 60;
* aged between 5 to 8 years.
* Inclusion in the experimental group was based on parents' motivation to follow such a heavy protocol both at home and for the one session per week at the hospital.
* Controls were matched for sex, age, IQ, study sites and treatment.

Exclusion Criteria:

* known organic syndrome and/or non-stabilized neuropediatric (e.g. seizures) or medical (e.g. diabetes mellitus) comorbidities.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
change from baseline in Autism Diagnostic Observation Schedule (ADOS) at 6 months | at baseline and 6 months

SECONDARY OUTCOMES:
change from baseline in Vineland II at 6 months | at baseline and 6 months
change from baseline in Child Behavior Check List at 6 months | at baseline and 6 months
change from baseline in Wechsler Intelligence scale at 6 months | at baseline and 6 months
change from baseline in Social Communication Questionnaire at 6 months | at baseline and 6 months
change from baseline in Parental Stress Index at 6 months | at baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Cohen, MD, PhD, Principal Investigator — Groupe hospitalier Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Derived] Jouen AL, Narzisi A, Xavier J, Tilmont E, Bodeau N, Bono V, Ketem-Premel N, Anzalone S, Maharatna K, Chetouani M, Muratori F, Cohen D; MICHELANGELO Study Group. GOLIAH (Gaming Open Library for Intervention in Autism at Home): a 6-month single blind matched controlled exploratory study. Child Adolesc Psychiatry Ment Health. 2017 Mar 22;11:17. doi: 10.1186/s13034-017-0154-7. eCollection 2017. PMID 28344643
- [Derived] Bono V, Narzisi A, Jouen AL, Tilmont E, Hommel S, Jamal W, Xavier J, Billeci L, Maharatna K, Wald M, Chetouani M, Cohen D, Muratori F; MICHELANGELO Study Group. GOLIAH: A Gaming Platform for Home-Based Intervention in Autism - Principles and Design. Front Psychiatry. 2016 Apr 28;7:70. doi: 10.3389/fpsyt.2016.00070. eCollection 2016. PMID 27199777